CLINICAL TRIAL: NCT04712110
Title: A Phase 1/2, Randomized, Observer-Blind, Placebo-Controlled Trial to Evaluate the Safety and Immunogenicity of TAK-019 by Intramuscular Injection in Healthy Japanese Male and Female Adults Aged 20 Years and Older (COVID-19)
Brief Title: A Study of TAK-019 in Healthy Japanese Adults (COVID-19)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TAK-019-1501; U1111-1262-6244 (Other: WHO); jRCT2071200084 (Registry Identifier: jRCT)
Record Dates: First submitted 2021-01-14; First posted 2021-01-15 (Actual); Results first posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: Prevention of Infection Disease Caused by Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- TAK-019 (Experimental): TAK-019 0.5 mL, intramuscular injection in the upper arm
  Interventions: Biological: TAK-019
- Placebo (Placebo Comparator): TAK-019 Matching Placebo, intramuscular injection in the upper arm
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: TAK-019 — TAK-019 intramuscular injection
  Arms: TAK-019
Biological: Placebo — Placebo intramuscular injection
  Arms: Placebo

SUMMARY:
TAK-019 is a vaccine in development to protect people against Covid-19. The main aims of the study are to learn if TAK-019 can protect people from Covid-19 and to check for side effects from TAK-019.

At the first visit, the study doctor will check if each person can take part. Those who can take part will be chosen for 1 of 2 treatments by chance. Participants will either receive an injection of TAK-019 or a placebo in their arm. In this study, a placebo will look like the TAK-019 vaccine but will not have any medicine in it. 3 times as many participants will receive TAK-019 than placebo. Participants will receive 2 injections of TAK-019 or placebo, 21 days apart.

Participants will be asked to record their temperature and any medical problems in an electronic diary for up to 7 days after each injection.

During the study, participants will visit the clinic for regular check-ups, blood tests, and sometimes for nose swab samples. When all participants have attended a clinic visit 28 days after their 2nd injection, the study sponsor (Takeda) will check how many participants have made enough antibodies to protect them against Covid-19.

The participants will stay in the study for up to 12 months after they have had their 2nd injection. During this time, the study doctors will continue to check how many participants have made enough antibodies to protect them against Covid-19. Also, they will check if participants have any more side effects from TAK-019 or the placebo.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-019. TAK-019 is being tested to prevent infectious disease caused by Severe Acute Respiratory Syndrome coronavirus-2 (SARS-CoV-2). This study will look at the evaluate the safety and immunogenicity of 2 doses of TAK-019 by intramuscular (IM) injection 21 days apart in healthy Japanese male and female adults.

The study will enroll approximately 200 healthy volunteers. Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups-which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* TAK-019 0.5 mL
* Placebo- this is an injection that looks like the study drug but has no active ingredient

All participants will be asked to take intramuscular injection in the upper arm twice throughout the study.

This multi-center trial will be conducted in Japan. The overall time to participate in this study is 12 months from the second vaccination (totally 387 days). Participants will make multiple visits to the clinic and will be contacted by telephone or a final visit after the last vaccination for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Japanese male and female adult participants aged >= 20 years of age at the time of signing of informed consent.
2. Participants who understand and are willing to comply with trial procedures and are available for the duration of follow-up.

Exclusion Criteria:

1. Participants who received any other SARS-CoV-2 or other experimental novel coronavirus vaccine prior to the trial.
2. Participants who have close contact of anyone known to have COVID-19 within 30 days prior to the trial vaccination.
3. Participants who were tested positive for SARS-CoV-2 prior to the trial or before the trial vaccination.
4. Participants who are on current treatment with other investigational agents for prophylaxis of COVID-19.
5. Participants who have traveled outside of Japan in the 30 days prior to the trial participation.
6. Participants with a clinically significant active infection (as assessed by the Investigator) or oral temperature >= 38 degree Celsius within 3 days of the intended date of vaccination.
7. Participants with known hypersensitivity or allergy to any of the investigational vaccine components.
8. Participants with history or any illness that, in the opinion of the Investigator, might interfere with the results of the trial or pose additional risk to the participants due to participation in the trial.
9. Participants with known or suspected impairment/alteration of immune function, including history of any autoimmune disease or neuro-inflammatory disease.
10. Abnormalities of splenic or thymic function.
11. Participants with a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.
12. Participants with any serious chronic or progressive disease (eg, neoplasm, insulin dependent diabetes, cardiac, renal or hepatic disease).
13. Participants with body mass index (BMI) greater than or equal to 30 kg/m^2 (BMI= weight in kg/ height in meters^2).
14. Participants participating in any clinical trial with another investigational product within 30 days prior to the trial vaccination or intend to participate in another clinical trial at any time during the conduct of this trial.
15. Participants who received or plan to receive any other licensed vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to trial dose administration.
16. Participants with acute or chronic clinically significant disease including pulmonary, cardiovascular, hepatic or renal abnormality evaluated by physical examination.
17. Participants involved in the trial conduct or their first degree relatives.
18. Participants who have history or infection of hepatitis B, hepatitis C, and human immunodeficiency virus infection.
19. Female participants who are pregnant or breastfeeding.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (2):
- Japan (2):
  - Sumida Hospital, Sumida-ku, Tokyo
  - Nishi Kumamoto Hospital, Kumamoto

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Masuda T, Murakami K, Sugiura K, Sakui S, Schuring RP, Mori M. Safety and immunogenicity of NVX-CoV2373 (TAK-019) vaccine in healthy Japanese adults: Interim report of a phase I/II randomized controlled trial. Vaccine. 2022 May 26;40(24):3380-3388. doi: 10.1016/j.vaccine.2022.04.035. Epub 2022 Apr 29. PMID 35501178
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/60084996565ce300294c6ad7

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in Japan from 12 February 2021 to 28 March 2022.
Pre-assignment Details: Healthy Japanese participants were enrolled to receive two doses of TAK-019 or placebo by intramuscular injection on Day 1 (first vaccination) and Day 22 (second vaccination).
Groups:
- Placebo: TAK-019 placebo-matching, injection, intramuscularly once on Days 1 and 22 in the healthy participants.
- TAK-019 0.5 mL: TAK-019 0.5 milliliter (mL), injection, intramuscularly, once on Days 1 and 22 in the healthy participants.
Period: Overall Study
Arm/Group | Placebo | TAK-019 0.5 mL
Started | 50 | 150
Completed | 4 | 131
Not Completed | 46 | 19
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Chose Publicly Available SARS-CoV-2 Vaccine | 46 | 14

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received at least 1 dose of the treatment.
Groups:
- TAK-019 0.5 mL: TAK-019 0.5 mL, injection, intramuscularly, once on Days 1 and 22 in the healthy participants.
- Total: Total of all reporting groups
Arm/Group | Placebo | TAK-019 0.5 mL | Total
Number analyzed (Participants) | 50 | 150 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (16.42) | 52.6 (15.80) | 52.2 (15.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 65 | 86
  Male | 29 | 85 | 114
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 50 | 150 | 200
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 50 | 150 | 200
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 61.73 (11.806) | 62.94 (10.485) | 62.64 (10.813)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 164.00 (9.157) | 164.10 (8.596) | 164.08 (8.716)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 22.80 (2.865) | 23.29 (2.850) | 23.17 (2.854)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Solicited Local Adverse Events (AEs) for Six Subsequent Days Following First Vaccination
Description: Solicited local AEs were pre-defined local (at the injection site) AEs for which participants were specifically questioned and which were noted by participants in their diary for six subsequent days following first vaccination. Solicited local AEs included injection site pain, tenderness, erythema/redness, induration, and swelling.
Time Frame: Up to Day 7 (6 subsequent days after first vaccination on Day 1)
Population: The safety analysis set included all participants who received at least 1 dose of the treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-019 0.5 mL
Number analyzed (Participants) | 50 | 150
percentage of participants
  Injection site pain | 4.0 | 29.3
  Tenderness | 4.0 | 43.3
  Erythema/redness | 0.0 | 2.7
  Induration | 0.0 | 3.3
  Swelling | 0.0 | 2.7

2. Primary Outcome: Percentage of Participants With Solicited Local AEs for Six Subsequent Days Following Second Vaccination
Description: Solicited local AEs were pre-defined local (at the injection site) AEs for which participants were specifically questioned and which were noted by participants in their diary for six subsequent days following second vaccination. Solicited local AEs included injection site pain, tenderness, erythema/redness, induration, and swelling.
Time Frame: Up to Day 28 (6 subsequent days after second vaccination on Day 22)
Population: The safety analysis set included all participants who received at least 1 dose of the treatment. Here, "overall number of participants analyzed" signifies those participants who received second vaccination.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-019 0.5 mL
Number analyzed (Participants) | 49 | 150
percentage of participants
  Injection site pain | 2.0 | 50.0
  Tenderness | 4.1 | 62.7
  Erythema/redness | 0.0 | 15.3
  Induration | 0.0 | 11.3
  Swelling | 0.0 | 17.3

3. Primary Outcome: Percentage of Participants With Solicited Systemic AEs for Six Subsequent Days Following First Vaccination
Description: Solicited systemic AEs were pre-defined AEs for which participants were specifically questioned and which were noted by participants in their diary for six subsequent days following first vaccination. Solicited systemic AEs included fever, fatigue, malaise, myalgia, arthralgia, nausea/vomiting and headache.
Time Frame: Up to Day 7 (6 subsequent days after first vaccination on Day 1)
Population: The safety analysis set included all participants who received at least 1 dose of the treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-019 0.5 mL
Number analyzed (Participants) | 50 | 150
percentage of participants
  Fever | 0.0 | 0.0
  Fatigue | 6.0 | 8.7
  Malaise | 4.0 | 10.0
  Myalgia | 4.0 | 17.3
  Arthralgia | 0.0 | 4.7
  Nausea/vomiting | 0.0 | 0.7
  Headache | 2.0 | 10.7

4. Primary Outcome: Percentage of Participants With Solicited Systemic AEs for Six Subsequent Days Following Second Vaccination
Description: Solicited systemic AEs were pre-defined AEs for which participants were specifically questioned and which were noted by participants in their diary for six subsequent days following second vaccination. Solicited systemic AEs included fever, fatigue, malaise, myalgia, arthralgia, nausea/vomiting and headache.
Time Frame: Up to Day 28 (6 subsequent days after second vaccination on Day 22)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-019 0.5 mL
Number analyzed (Participants) | 49 | 150
percentage of participants
  Fever | 0.0 | 6.0
  Fatigue | 8.2 | 20.7
  Malaise | 6.1 | 29.3
  Myalgia | 4.1 | 32.7
  Arthralgia | 0.0 | 13.3
  Nausea/vomiting | 0.0 | 5.3
  Headache | 2.0 | 21.3

5. Primary Outcome: Percentage of Participants With Unsolicited AEs for 20 Days Following First Vaccination
Description: Unsolicited AEs were all AEs that were not pre-defined for which the participant was not specifically questioned in the participant diary.
Time Frame: Up to Day 21 (20 days after first vaccination on Day 1)
Population: The safety analysis set included all participants who received at least 1 dose of the treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-019 0.5 mL
Number analyzed (Participants) | 50 | 150
percentage of participants | 8.0 | 10.0

6. Primary Outcome: Percentage of Participants With Unsolicited AEs for 27 Days Following Second Vaccination
Description: as for outcome 5
Time Frame: Up to Day 49 (27 days after second vaccination on Day 22)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-019 0.5 mL
Number analyzed (Participants) | 49 | 150
percentage of participants | 12.2 | 29.3

7. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) Until Day 50
Description: Only unsolicited SAEs data was planned to be collected and assessed for the assessment of this outcome measure (OM) and solicited SAE was out of the scope of assessment. Unsolicited SAEs were those AEs that were not pre-defined for which the participant was not specifically questioned in the participant diary. Percentage of participants with unsolicited SAEs until Day 50 were reported in this outcome measure.
Time Frame: Day 1 up to Day 50
Population: The safety analysis set included all participants who received at least 1 dose of the treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-019 0.5 mL
Number analyzed (Participants) | 50 | 150
percentage of participants | 0.0 | 0.0

8. Primary Outcome: Percentage of Participants With Adverse Events of Special Interest (AESI) Until Day 50
Description: AESIs were defined as AEs that were specifically highlighted to the Investigator. Only unsolicited AESI data was planned to be collected and assessed for the assessment of this OM and solicited AESI was out of the scope of assessment. Unsolicited AESIs were those AEs that were not pre-defined for which the participant was not specifically questioned in the participant diary. Percentage of participants with unsolicited AESIs until Day 50 were reported in this outcome measure.
Time Frame: Day 1 up to Day 50
Population: The safety analysis set included all participants who received at least 1 dose of the treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-019 0.5 mL
Number analyzed (Participants) | 50 | 150
percentage of participants | 0.0 | 0.0

9. Primary Outcome: Percentage of Participants With Medically-Attended Adverse Events (MAAEs) Until Day 50
Description: MAAEs are defined as AEs leading to an unscheduled visit to or by a healthcare professional including visits to an emergency department, but not fulfilling seriousness criteria. Only unsolicited MAAEs data was planned to be collected and assessed for the assessment of this OM and solicited MAAE was out of the scope of assessment. Unsolicited MAAEs were those AEs that were not pre-defined for which the participant was not specifically questioned in the participant diary. Percentage of participants with unsolicited MAAEs until Day 50 were reported in this outcome measure.
Time Frame: Day 1 up to Day 50
Population: The safety analysis set included all participants who received at least 1 dose of the treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-019 0.5 mL
Number analyzed (Participants) | 50 | 150
percentage of participants | 4.0 | 2.7

10. Primary Outcome: Percentage of Participants With Any AE Leading to Discontinuation of Vaccination
Description: Only any unsolicited AE leading to discontinuation of vaccination data was planned to be collected and assessed for the assessment of this OM and solicited AE leading to discontinuation of vaccination was out of the scope of assessment. Unsolicited AEs were those AEs that were not pre-defined for which the participant was not specifically questioned in the participant diary. Percentage of participants with any unsolicited AE leading to discontinuation of vaccination until Day 22 were reported in this outcome measure.
Time Frame: Day 1 up to Day 22
Population: The safety analysis set included all participants who received at least 1 dose of the treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-019 0.5 mL
Number analyzed (Participants) | 50 | 150
percentage of participants | 2.0 | 0.0

11. Primary Outcome: Percentage of Participants With Any AE Leading to Participant's Withdrawal From the Trial Until Day 50
Description: Only any unsolicited AE leading to participant's withdrawal from the trial data was planned to be collected and assessed for the assessment of this OM and solicited AE leading to participant's withdrawal from the trial was out of the scope of assessment. Unsolicited AEs were those AEs that were not pre-defined for which the participant was not specifically questioned in the participant diary. Percentage of participants with any unsolicited AE leading to participant's withdrawal from the trial until Day 50 were reported in this outcome measure.
Time Frame: Day 1 up to Day 50
Population: The safety analysis set included all participants who received at least 1 dose of the treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-019 0.5 mL
Number analyzed (Participants) | 50 | 150
percentage of participants | 0.0 | 0.0

12. Primary Outcome: Percentage of Participants With Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) Infection Until Day 50
Time Frame: Day 1 up to Day 50
Population: The safety analysis set included all participants who received at least 1 dose of the treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-019 0.5 mL
Number analyzed (Participants) | 50 | 150
percentage of participants | 0.0 | 0.0

13. Primary Outcome: Geometric Mean Titers (GMT) of Serum Immunoglobulin G (IgG) Antibody Levels to SARS-CoV-2 Recombinant Spike (rS) Protein on Day 36
Description: GMT was the immunogenicity outcome expressed as reciprocal antibody titer with average for each group. Titer values was measured as below lower limit of quantification (LLOQ) were imputed to a value that was half of the LLOQ. LLOQ was equal to 200. Here, ELISA is Enzyme-linked immunosorbent assay.
Time Frame: At Day 36
Population: The per-protocol set (PPS) included all randomized participants who received at least one dose of treatment and had evaluable immunogenicity data and did not have significant protocol deviations which influenced the immunogenicity assessment.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units per mL (EU/mL)
Arm/Group | Placebo | TAK-019 0.5 mL
Number analyzed (Participants) | 49 | 150
ELISA units per mL (EU/mL) | 132.3 [109.6 to 159.5] | 31036.8 [26837.1 to 35893.7]

14. Primary Outcome: Geometric Mean Fold Rise (GMFR) of Serum IgG Antibody Levels to SARS-CoV-2 rS Protein on Day 36
Description: GMFR was calculated as the ratio of the post-vaccination titer level to the baseline titer level. Baseline was defined as the last measurement taken before the first dose of study intervention.
Time Frame: At Day 36
Population: The PPS included all randomized participants who received at least one dose of treatment and had evaluable immunogenicity data and did not have significant protocol deviations which influenced the immunogenicity assessment.
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Placebo | TAK-019 0.5 mL
Number analyzed (Participants) | 49 | 150
fold change | 1.0 [1.0 to 1.1] | 258.8 [218.8 to 306.0]

15. Primary Outcome: Seroconversion Rate (SCR) of Serum IgG Antibody Levels to SARS-CoV-2 rS Protein on Day 36
Description: SCR was defined as percentage of participants with 4-fold or more rises in titer if naive at baseline OR percentage of participants with 2-fold or more rises in titer if seropositive at baseline. Baseline was defined as the last measurement taken before the first dose of study intervention.
Time Frame: At Day 36
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | TAK-019 0.5 mL
Number analyzed (Participants) | 49 | 150
percentage of participants | 0.0 [0.0 to 7.3] | 100.0 [97.6 to 100.0]

16. Primary Outcome: Seroresponse Rate (SRR) of Serum IgG Antibody Levels to SARS-CoV-2 rS Protein on Day 36
Description: SRR was defined as percentage of participants with greater than or equal to (>=) 95 percentile in titer at Baseline for all participants. Baseline was defined as the last measurement taken before the first dose of study intervention.
Time Frame: At Day 36
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | TAK-019 0.5 mL
Number analyzed (Participants) | 49 | 150
percentage of participants | 8.2 [2.3 to 19.6] | 100.0 [97.6 to 100.0]

17. Secondary Outcome: Percentage of Participants With SAE Throughout the Trial
Description: Only unsolicited SAEs data was planned to be collected and assessed for the assessment of this OM and solicited SAE was out of the scope of assessment. Unsolicited SAEs were those AEs that were not pre-defined for which the participant was not specifically questioned in the participant diary. Percentage of participants with unsolicited SAEs throughout the trial were reported in this outcome measure.
Time Frame: Day 1 up to Day 387
Population: The safety analysis set included all participants who received at least 1 dose of the treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-019 0.5 mL
Number analyzed (Participants) | 50 | 150
percentage of participants | 2.0 | 0.0

18. Secondary Outcome: Percentage of Participants With AESI Throughout the Trial
Description: AESIs were defined as AEs that were specifically highlighted to the Investigator. Only unsolicited AESI data was planned to be collected and assessed for the assessment of this OM and solicited AESI was out of the scope of assessment. Unsolicited AESI were those AEs that were not pre-defined for which the participant was not specifically questioned in the participant diary. Percentage of participants with unsolicited AESIs throughout the trial were reported in this outcome measure.
Time Frame: Day 1 up to Day 387
Population: The safety analysis set included all participants who received at least 1 dose of the treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-019 0.5 mL
Number analyzed (Participants) | 50 | 150
percentage of participants | 0.0 | 0.0

19. Secondary Outcome: Percentage of Participants With MAAEs Throughout the Trial
Description: MAAEs are defined as AEs leading to an unscheduled visit to or by a healthcare professional including visits to an emergency department, but not fulfilling seriousness criteria. Only unsolicited MAAEs data was planned to be collected and assessed for the assessment of this OM and solicited MAAE was out of the scope of assessment. Unsolicited MAAEs were those AEs that were not pre-defined for which the participant was not specifically questioned in the participant diary. Percentage of participants with unsolicited MAAEs throughout the trial were reported in this outcome measure.
Time Frame: Day 1 up to Day 387
Population: The safety analysis set included all participants who received at least 1 dose of the treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-019 0.5 mL
Number analyzed (Participants) | 50 | 150
percentage of participants | 6.0 | 10.7

20. Secondary Outcome: Percentage of Participants With Any AE Leading to Participant's Withdrawal From the Trial From the Day of Vaccination Throughout the Trial
Description: Only any unsolicited AE leading to participant's withdrawal from the trial data was planned to be collected and assessed for the assessment of this OM and solicited AE leading to participant's withdrawal from the trial was out of the scope of assessment. Unsolicited AEs were those AEs that were not pre-defined for which the participant was not specifically questioned in the participant diary. Percentage of participants with any unsolicited AE leading to withdrawal from the trial from the day of vaccination throughout the trial were reported in this outcome measure.
Time Frame: Day 1 up to Day 387
Population: The safety analysis set included all participants who received at least 1 dose of the treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-019 0.5 mL
Number analyzed (Participants) | 50 | 150
percentage of participants | 0.0 | 0.0

21. Secondary Outcome: Percentage of Participants With SARS-CoV-2 Infection Throughout the Trial
Time Frame: Day 1 up to Day 387
Population: The safety analysis set included all participants who received at least 1 dose of the treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-019 0.5 mL
Number analyzed (Participants) | 50 | 150
percentage of participants | 2.0 | 2.7

22. Secondary Outcome: GMT of Serum IgG Antibody Levels to SARS-CoV-2 rS Protein on Days 22, 50, 202, and 387
Description: GMT was the immunogenicity outcome expressed as reciprocal antibody titer with average for each group. Titer values was measured as below LLOQ were imputed to a value that was half of the LLOQ. GMT of serum IgG antibody levels to the SARS-CoV-2 rS protein was measured where LLOQ was equal to 200.
Time Frame: At Days 22, 50, 202, and 387
Population: The PPS included all randomized participants who received at least one dose of treatment and had evaluable immunogenicity data and did not have significant protocol deviations which influenced the immunogenicity assessment. Here, "number analyzed" signifies those participants who were evaluable for this outcome measure at given timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Placebo | TAK-019 0.5 mL
Number analyzed (Participants) | 49 | 150
EU/mL
  Day 22 | 144.9 [115.2 to 182.4] | 1390.0 [1140.8 to 1693.7]
  Day 50: number analyzed (Participants) | 49 | 149
  Day 50 | 134.7 [109.3 to 166.2] | 23910.8 [20737.0 to 27570.3]
  Day 202: number analyzed (Participants) | 6 | 146
  Day 202 | 851.0 [26.0 to 27800.8] | 4390.1 [3600.9 to 5352.3]
  Day 387: number analyzed (Participants) | 4 | 127
  Day 387 | 236.7 [15.2 to 3674.6] | 3461.2 [2601.5 to 4605.1]

23. Secondary Outcome: GMFR of Serum IgG Antibody Levels to SARS-CoV-2 rS Protein on Days 22, 50, 202, and 387
Description: GMFR was calculated as the ratio of the post-vaccination titer level to the baseline titer level. Where baseline was defined as the last measurement taken before the first dose of study intervention.
Time Frame: At Days 22, 50, 202, and 387
Population: as for outcome 22
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Placebo | TAK-019 0.5 mL
Number analyzed (Participants) | 49 | 150
fold change
  Day 22 | 1.1 [1.0 to 1.2] | 11.6 [9.4 to 14.2]
  Day 50: number analyzed (Participants) | 49 | 149
  Day 50 | 1.0 [1.0 to 1.1] | 199.1 [169.2 to 234.3]
  Day 202: number analyzed (Participants) | 6 | 146
  Day 202 | 8.5 [0.3 to 278.0] | 36.4 [29.8 to 44.6]
  Day 387: number analyzed (Participants) | 4 | 127
  Day 387 | 2.4 [0.2 to 36.7] | 27.9 [20.7 to 37.6]

24. Secondary Outcome: SCR of Serum IgG Antibody Levels to SARS-CoV-2 rS Protein on Days 22, 50, 202, and 387
Description: as for outcome 15
Time Frame: At Days 22, 50, 202, and 387
Population: as for outcome 22
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | TAK-019 0.5 mL
Number analyzed (Participants) | 49 | 150
percentage of participants
  Day 22 | 6.1 [1.3 to 16.9] | 82.7 [75.6 to 88.4]
  Day 50: number analyzed (Participants) | 49 | 149
  Day 50 | 2.0 [0.1 to 10.9] | 100.0 [97.6 to 100.0]
  Day 202: number analyzed (Participants) | 6 | 146
  Day 202 | 33.3 [4.3 to 77.7] | 97.9 [94.1 to 99.6]
  Day 387: number analyzed (Participants) | 4 | 127
  Day 387 | 25.0 [0.6 to 80.6] | 96.9 [92.1 to 99.1]

25. Secondary Outcome: SRR of Serum IgG Antibody Levels to SARS-CoV-2 rS Protein on Days 22, 50, 202, and 387
Description: SRR was defined as percentage of participants with >=95 percentile in titer at Baseline for all participants. Baseline was defined as the last measurement taken before the first dose of study intervention.
Time Frame: At Days 22, 50, 202, and 387
Population: as for outcome 22
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | TAK-019 0.5 mL
Number analyzed (Participants) | 49 | 150
percentage of participants
  Day 22 | 10.2 [3.4 to 22.2] | 84.0 [77.1 to 89.5]
  Day 50: number analyzed (Participants) | 49 | 149
  Day 50 | 12.2 [4.6 to 24.8] | 100.0 [97.6 to 100.0]
  Day 202: number analyzed (Participants) | 6 | 146
  Day 202 | 33.3 [4.3 to 77.7] | 97.9 [94.1 to 99.6]
  Day 387: number analyzed (Participants) | 4 | 127
  Day 387 | 25.0 [0.6 to 80.6] | 96.9 [92.1 to 99.1]

26. Secondary Outcome: GMT of Serum Neutralizing Antibody (nAb) Titers to Wild Type Virus on Days 22, 36, 50, 202 and Day 387
Description: The neutralization titer was expressed as the reciprocal of the highest dilution at which greater than or equal to (>=) 50% of the replicate wells were protected from infection (MN50). GMT was the immunogenicity outcome expressed as reciprocal antibody titer with average for each group. Titer values was measured as below LLOQ were imputed to a value that was half of the LLOQ. GMT of serum IgG antibody levels to the SARS-CoV-2 rS protein was measured where LLOQ was equal to 20.
Time Frame: At Days 22, 36, 50, 202 and 387
Population: as for outcome 22
Measure: Geometric Mean (95% Confidence Interval); unit: 1 per dilution
Arm/Group | Placebo | TAK-019 0.5 mL
Number analyzed (Participants) | 49 | 150
1 per dilution
  Day 22 | 10.4 [9.9 to 10.9] | 50.2 [41.2 to 61.0]
  Day 36 | 10.4 [9.9 to 10.9] | 884.4 [749.0 to 1044.4]
  Day 50: number analyzed (Participants) | 49 | 149
  Day 50 | 10.4 [9.9 to 10.9] | 509.5 [422.5 to 614.6]
  Day 202: number analyzed (Participants) | 6 | 146
  Day 202 | 50.4 [3.6 to 698.8] | 65.5 [53.4 to 80.4]
  Day 387: number analyzed (Participants) | 4 | 127
  Day 387 | 14.1 [4.7 to 42.6] | 65.7 [49.0 to 88.1]

27. Secondary Outcome: GMFR of Serum nAb Titers to Wild Type Virus on Days 22, 36, 50, 202 and 387
Description: The neutralization titer was expressed as the reciprocal of the highest dilution at which >=50% of the replicate wells were protected from infection (MN50). GMFR was calculated as the ratio of the post-vaccination titer level to the baseline titer level. Baseline was defined as the last measurement taken before the first dose of study intervention.
Time Frame: At Days 22, 36, 50, 202 and 387
Population: as for outcome 22
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | Placebo | TAK-019 0.5 mL
Number analyzed (Participants) | 49 | 150
fold change
  Day 22 | 1.0 [1.0 to 1.1] | 5.0 [4.1 to 6.1]
  Day 36 | 1.0 [1.0 to 1.1] | 88.0 [74.5 to 104.0]
  Day 50: number analyzed (Participants) | 49 | 149
  Day 50 | 1.0 [1.0 to 1.1] | 50.7 [42.0 to 61.2]
  Day 202: number analyzed (Participants) | 6 | 146
  Day 202 | 5.0 [0.4 to 69.9] | 6.5 [5.3 to 8.0]
  Day 387: number analyzed (Participants) | 4 | 127
  Day 387 | 1.4 [0.5 to 4.3] | 6.5 [4.9 to 8.7]

28. Secondary Outcome: SCR to Serum nAb Titers to Wild Type Virus on Days 22, 36, 50, 202 and 387
Description: The neutralization titer was expressed as the reciprocal of the highest dilution at which >=50% of the replicate wells were protected from infection (MN50). SCR was defined as percentage of participants with 4-fold or more rises in titer if naive at baseline OR percentage of participants with 2-fold or more rises in titer if seropositive at Baseline. Baseline was defined as the last measurement taken before the first dose of study intervention.
Time Frame: At Days 22, 36, 50, 202 and 387
Population: as for outcome 22
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | TAK-019 0.5 mL
Number analyzed (Participants) | 49 | 150
percentage of participants
  Day 22 | 0.0 [0.0 to 7.3] | 67.3 [59.2 to 74.8]
  Day 36 | 0.0 [0.0 to 7.3] | 99.3 [96.3 to 100.0]
  Day 50: number analyzed (Participants) | 49 | 149
  Day 50 | 0.0 [0.0 to 7.3] | 98.0 [94.2 to 99.6]
  Day 202: number analyzed (Participants) | 6 | 146
  Day 202 | 33.3 [4.3 to 77.7] | 76.0 [68.3 to 82.7]
  Day 387: number analyzed (Participants) | 4 | 127
  Day 387 | 25.0 [0.6 to 80.6] | 70.9 [62.1 to 78.6]

29. Secondary Outcome: SRR to Serum nAb Titers to Wild Type Virus on Days 22, 36, 50, 202 and 387
Description: The neutralization titer was expressed as the reciprocal of the highest dilution at which >=50% of the replicate wells were protected from infection (MN50). SRR was defined as percentage of participants with >=95 percentile in titer at Baseline for all participants. Baseline was defined as the last measurement taken before the first dose of study intervention.
Time Frame: At Days 22, 36, 50, 202 and 387
Population: as for outcome 22
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | TAK-019 0.5 mL
Number analyzed (Participants) | 49 | 150
percentage of participants
  Day 22 | 100.0 [92.7 to 100.0] | 100.0 [97.6 to 100.0]
  Day 36 | 100.0 [92.7 to 100.0] | 100.0 [97.6 to 100.0]
  Day 50: number analyzed (Participants) | 49 | 149
  Day 50 | 100.0 [92.7 to 100.0] | 100.0 [97.6 to 100.0]
  Day 202: number analyzed (Participants) | 6 | 146
  Day 202 | 100.0 [54.1 to 100.0] | 100.0 [97.5 to 100.0]
  Day 387: number analyzed (Participants) | 4 | 127
  Day 387 | 100.0 [39.8 to 100.0] | 100.0 [97.1 to 100.0]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) are AEs that started after the first vaccination on Day 1 up to 365 days after the second vaccination on Day 22 (Day 387)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Groups:
- TAK-019: TAK-019 0.5 mL, injection, intramuscularly, once on Days 1 and 22 in the healthy participants.
Arm/Group | Placebo | TAK-019
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/150
Serious Adverse Events (participants affected / at risk) | 1/50 | 0/150
Other Adverse Events (participants affected / at risk) | 11/50 | 124/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=50) | TAK-019 (N=150)
COVID-19 (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=50) | TAK-019 (N=150)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 24
Body temperature increased (Investigations) | 0 | 9
Fatigue (General disorders) | 7 | 39
Headache (Nervous system disorders) | 2 | 41
Induration (General disorders) | 0 | 20
Injection site pain (General disorders) | 3 | 88
Injection site pruritus (General disorders) | 0 | 26
Malaise (General disorders) | 6 | 50
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 56
Nausea (Gastrointestinal disorders) | 0 | 9
Swelling (General disorders) | 0 | 27
Tenderness (General disorders) | 3 | 100
Vaccination site erythema (General disorders) | 0 | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2021-04-09): https://cdn.clinicaltrials.gov/large-docs/10/NCT04712110/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/10/NCT04712110/SAP_001.pdf